CLINICAL TRIAL: NCT04831970
Title: POst-Prostatectomy Ablative Radiation Therapy
Acronym: POPART
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Stefano Arcangeli, Associate Professor, University of Milano Bicocca
Other Study IDs: POPART
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Radiation Toxicity
Keywords: SBRT; adjuvant RT; salvage RT; prostatectomy; prostatic bed
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of hypofractionated radiotherapy for prostate cancer has matured to a point that in current guidelines extremely hypofractionated image-guided IMRT regimens (6 Gy per fraction or greater) can be considered an alternative to conventionally fractionated regimens at clinics with appropriate technology, physics and clinical expertise. The delivery of fewer and larger fractions with hypofractionation compared to conventional radiotherapy might effectively improve the therapeutic ratio while maintaining isoeffective tumour doses, thus, shortening overall treatment time. In the present study, patients will undergo postoperative image-guided SBRT by means of volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) with state-of-the-art treatment-planning and quality assurance procedures. Normal tissue sparing and delivery accuracy are accomplished by the use of devices that ensure stability and beam location reproducibility. The primary endpoint is to evaluate the cumulative incidence of treatment related toxicities and adverse events in the acute (< 90 days from the end of treatment) and late (> 90 days) setting.

DETAILED DESCRIPTION:
In this observational prospective trial eligible patients are those with adverse pathological features or rising PSA after radical prostatectomy proposed for receiving 31 Gy in 5 sessions each of 6.2 Gy to the prostatic bed delivered in one week, and up to 32.5 Gy in 5 sessions each of 6.5 Gy delivered in one week, respectively, in case of clinical relapse.

Patients will be treated by means of image guided volumetric modulated radiotherapy (IGRT-VMAT). A real time non-ionizing target monitoring might be used to account for intra-fractional errors, if deemed appropriate. Whether the dose constraints to the normal tissues are at risk, these will be prioritised over the prescription dose to the target. The primary endpoint of the trial is to assess the treatment related toxicity measured by the CTCAE v5.0. Secondary endpoints are quality of life in different domains (sexual, rectal , urinary) and biochemical outcome.

Patients will be followed at approximately one month, then every 3 months for the first 12 months and every 6 months thereafter. Quality of Life will be prospectively evaluated through validated tools (ECOG, EPIC, IIEF-5, ICIQ-SF) at various timepoints. Percentage or total mean score will be reported according to the questionnaires, whether they grade values in a scale or use descriptive statistics. Kaplan-Meier curve analysis of biochemical relapse free survival (b-RFS) at 2 and 5-year bRFS for all patients will be estimated.

ELIGIBILITY:
INCLUSION CRITERIA

* Adenocarcinoma of the prostate treated with radical prostatectomy (any type of radical prostatectomy is permitted including retropubic, perineal, laparoscopic or robotically assisted; there is no time limit for the date of radical prostatectomy).
* Pathologic T3N0/Nx disease or pathologic T2N0/Nx disease, with or without a positive prostatectomy surgical margin
* Post-radical prostatectomy PSA of ≥ 0.1 - < 2.0 ng/mL.
* Clinical local relapse assessed by Magnetic Resonance Imaging (MRI) of the pelvis
* ECOG performance status of 0-1
* No distant metastases at restaging (in case of biochemical failure), within 60 days prior to registration
* Patients can be on androgen deprivation therapy
* Ability to understand and willingness to sign a study-specific informed consent prior to study entry

EXCLUSION CRITERIA

* N1 and or M1 patients
* Prior radiation of any kind to the prostate gland or pelvis
* Prior brachytherapy is not allowed
* History of inflammatory colitis or other active severe comorbidities
* Patients who are on immunosuppressant medication

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adverse pathological features or biochemical and clinical relapse following radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v.5.0 | 60 months
  To assess treatment related acute (< 90 days from the end of treatment) and late (> 90 days) gastrointestinal (GI) and genitourinary (GU) toxicity in patients who undergo postoperative SBRT using CTCAE v.5.0

SECONDARY OUTCOMES:
QUALITY OF LIFE (QOL) assessed by Expanded Prostate Cancer Index Composite (EPIC-26) Questionnaire. For each domain minimum symptom score (=0) means best QOL and maximum symptom score (=12) means worst QOL | 60 months
  To measure symptom scores for each QOL domain (urinary incontinence, urinary irritative/obstructive, bowel, sexual) after SDRT by EPIC-26 Questionnaire
Number of participants with urinary incontinence assessed by International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), ranging from 0 (best) to 21 (worst) | 60 months
  To assess urinary continence after postoperative SBRT using ICIQ-SF
Number of participants with erectile dysfunction assessed by International Index of Erectile Function Questionnaire ranging from 5 (worst ) to 25 (best) | 60 months
  To assess erectile function after postoperative SBRT using IIEF 5
Number of participants with biochemical relapse assessed by PSA (cut off 0.20 ng/mL) | 60 months
  To assess biochemical outcome after postoperative SBRT using serum PSA levels

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Arcangeli, MD, Principal Investigator — University of Milan Bicocca
Locations (2):
- Italy (2):
  - Radiation Oncology, Humanitas Cancer Center (Humanitas University), Rozzano, MI
  - Radiation Oncology, ASST Monza (University of Milan Bicocca), Monza

IPD SHARING:
Plan to Share IPD: Yes
outcomes of individual participant data sets will be shared with other investigators involved in the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years

REFERENCES:
- [Result] Morgan SC, Hoffman K, Loblaw DA, Buyyounouski MK, Patton C, Barocas D, Bentzen S, Chang M, Efstathiou J, Greany P, Halvorsen P, Koontz BF, Lawton C, Leyrer CM, Lin D, Ray M, Sandler H. Hypofractionated Radiation Therapy for Localized Prostate Cancer: An ASTRO, ASCO, and AUA Evidence-Based Guideline. J Clin Oncol. 2018 Oct 11;36(34):JCO1801097. doi: 10.1200/JCO.18.01097. Online ahead of print. No abstract available. PMID 30307776
- [Result] Kruser TJ, Jarrard DF, Graf AK, Hedican SP, Paolone DR, Wegenke JD, Liu G, Geye HM, Ritter MA. Early hypofractionated salvage radiotherapy for postprostatectomy biochemical recurrence. Cancer. 2011 Jun 15;117(12):2629-36. doi: 10.1002/cncr.25824. Epub 2010 Dec 14. PMID 21656740
- [Result] Bell LJ, Eade T, Hruby G, Bromley R, Kneebone A. Intra-fraction displacement of the prostate bed during post-prostatectomy radiotherapy. Radiat Oncol. 2021 Jan 22;16(1):20. doi: 10.1186/s13014-020-01743-9. PMID 33482863
- [Result] Wong GW, Palazzi-Churas KL, Jarrard DF, Paolone DR, Graf AK, Hedican SP, Wegenke JD, Ritter MA. Salvage hypofractionated radiotherapy for biochemically recurrent prostate cancer after radical prostatectomy. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):449-55. doi: 10.1016/j.ijrobp.2007.06.042. Epub 2007 Sep 14. PMID 17869014
- [Result] Wages NA, Sanders JC, Smith A, Wood S, Anscher MS, Varhegyi N, Krupski TL, Harris TJ, Showalter TN. Hypofractionated Postprostatectomy Radiation Therapy for Prostate Cancer to Reduce Toxicity and Improve Patient Convenience: A Phase 1/2 Trial. Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1254-1262. doi: 10.1016/j.ijrobp.2020.11.009. Epub 2020 Nov 21. PMID 33227441
- [Result] Ballas LK, Luo C, Chung E, Kishan AU, Shuryak I, Quinn DI, Dorff T, Jhimlee S, Chiu R, Abreu A, Jennelle R, Aron M, Groshen S. Phase 1 Trial of SBRT to the Prostate Fossa After Prostatectomy. Int J Radiat Oncol Biol Phys. 2019 May 1;104(1):50-60. doi: 10.1016/j.ijrobp.2018.12.047. Epub 2018 Dec 31. PMID 30605751
- [Result] Cuccia F, Mortellaro G, Serretta V, Valenti V, Tripoli A, Gueci M, Luca N, Lo Casto A, Ferrera G. Hypofractionated postoperative helical tomotherapy in prostate cancer: a mono-institutional report of toxicity and clinical outcomes. Cancer Manag Res. 2018 Oct 29;10:5053-5060. doi: 10.2147/CMAR.S182016. eCollection 2018. PMID 30464605
- [Result] Lewis SL, Patel P, Song H, Freedland SJ, Bynum S, Oh D, Palta M, Yoo D, Oleson J, Salama JK. Image Guided Hypofractionated Postprostatectomy Intensity Modulated Radiation Therapy for Prostate Cancer. Int J Radiat Oncol Biol Phys. 2016 Mar 1;94(3):605-11. doi: 10.1016/j.ijrobp.2015.11.025. Epub 2015 Dec 2. PMID 26867889
- [Result] Koerber SA, Katayama S, Sander A, Jaekel C, Haefner MF, Debus J, Herfarth K. Prostate bed irradiation with alternative radio-oncological approaches (PAROS) - a prospective, multicenter and randomized phase III trial. Radiat Oncol. 2019 Jul 10;14(1):122. doi: 10.1186/s13014-019-1325-x. PMID 31291969
- [Derived] Lucchini R, Franzese C, Vukcaj S, Purrello G, Panizza D, Faccenda V, Andreoli S, Poli GL, Baldaccini D, Lo Faro L, Tomatis S, Cazzaniga LF, Scorsetti M, Arcangeli S. Acute Toxicity and Quality of Life in a Post-Prostatectomy Ablative Radiation Therapy (POPART) Multicentric Trial. Curr Oncol. 2022 Nov 30;29(12):9349-9356. doi: 10.3390/curroncol29120733. PMID 36547147